CLINICAL TRIAL: NCT03579628
Title: An Open-label, Dose-escalation Phase I/Ib Study to Assess the Safety, Pharmacokinetics and Pharmacodynamics of AsiDNA, a DNA Repair Inhibitor Administered Intravenously, as Single Agent and to Assess the Safety and the Efficacy of AsiDNA in Combination With Carboplatin With or Without Paclitaxel, in Patients With Advanced Solid Tumors
Brief Title: AsiDNA (a DNA Repair Inhibitor) Administered IntraVenously in Advanced Solid Tumors
Acronym: DRIIV-1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Valerio Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OX2016-203-01
Record Dates: First submitted 2018-04-06; First posted 2018-07-06 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Advanced Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AsiDNA (Experimental): Part A: AsiDNA as a single agent:
  The study will follow a dose escalation "3 + 3" cohort design (with 6 dose levels).
  All patients will receive a loading dose of AsiDNA for 3 consecutive days as iv infusion at Day 1 (D1), Day 2 (D2) and Day 3 (D3), followed by iv infusion once a week (at D8 and D15 of a 21 days treatment period (1 cycle = 21 days). Each subsequent cycle will be administered on a weekly basis (D1, D8, D15) of a 21 days treatment period.
  Part B: AsiDNA combination with Carboplatin with or without Paclitaxel (Background treatments):
  * Part B1: Combination cohort of AsiDNA at DL3 (600mg) with Carboplatin AUC 5.
  * Part B2: Combination cohort of AsiDNA at DL3 (600mg) with Carboplatin AUC 5 and weekly Paclitaxel: 80 mg/m2 (full dose).
  Interventions: Drug: AsiDNA

INTERVENTIONS:
Drug: AsiDNA — All patients will receive a loading dose of AsiDNA iv infusion (D1, D2, D3) followed by weekly iv administrations.
  At cycle 1: Part B1: Carboplatin will be administered by a 1 hour IV infusion at D8, 1 hour after the end of AsiDNA infusion. Part B2: Carboplatin will be administered by a 1 hour IV infusion at D8, 1 hour after the end of AsiDNA infusion and Paclitaxel will be administered by a 1 hour IV infusion at D8, D15, D22 or 1 hour after the end of AsiDNA infusion for weekly administrations.
  At each other cycle: AsiDNA will be administered on a weekly basis. Part B1: Carboplatin will be administered by a 1 hour IV infusion at D1, 1 hour after the end of AsiDNA infusion. Part B2; Carboplatin will be administered by a 1 hour IV infusion at D1, 1 hour after the end of AsiDNA infusion and Paclitaxel will be administered on a weekly basis by a 1 hour IV infusion.
  Patients will continue study treatment until disease progression, unacceptable toxicity or patient's refusal to continue.

SUMMARY:
The aim of the study is to assess:

* Part A: the safety, pharmacokinetics, pharmacodynamics and preliminary efficacy of AsiDNA in patients with advanced solid tumors.
* Part B: the safety and preliminary efficacy of AsiDNA in combination with Carboplatin with or without Paclitaxel in patients with Advanced solid tumors.

ELIGIBILITY:
Key Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Life expectancy of at least 3 months.
* Patient with histologically or cytologically documented advanced/metastatic primary or recurrent solid tumors who failed or are not eligible to standard therapy (Part A) and who are candidate to Carboplatin (Part B1) and to Carboplatin and Paclitaxel (Part B2).
* Part A: Fresh tumor sample from a biopsy
* Part B: A most recent available tumor sample from a biopsy for all patients will be collected for retrospective analysis of 6 genes expression profile for validation of further stratification approach (exploratory purpose).
* Prior anticancer therapies (chemotherapy, radiation therapy, hormonal therapy, immunotherapy, biological therapy) are allowed under conditions
* At least one measurable lesion according to RECIST 1.1; Patient with no measurable lesion can be enrolled, if the tumor evaluation can be properly documented
* Must meet select hematological and biochemical laboratory indices

Part B only:

* Patient must be eligible to Carboplatin (Part B1) and to Carboplatin + weekly Paclitaxel (Part B2).
* Patients must not have received more than 6 prior cycles of platinum-based chemotherapy.

Key Exclusion Criteria:

* Patient with symptomatic/active central nervous system (CNS) metastases
* Other tumor location necessitating an urgent therapeutic intervention
* Patient with uncontrolled disease-related metabolic disorder
* Patient presenting the following abnormal laboratory values at screening:

  1. hematuria > 1+ on dipstick,
  2. proteinuria > 1+ on dipstick
* Patient with uncontrolled congestive heart failure defined as New York Heart Association (NYHA) class III or IV, uncontrolled hypertension, unstable heart disease
* Patient with significant ECG abnormalities defined as any cardiac dysrhythmia (> grade 2)
* Patient with significant chronic liver disease or active HBV or HCV infection
* Patients with HIV infection or an active infection requiring specific anti-infective therapy
* Participation in another clinical trial with any investigational drug within 28 days prior to first study drug administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2018-04-05 (Actual); Primary Completion 2021-02-24 (Actual); Study Completion 2022-02-20 (Actual)

PRIMARY OUTCOMES:
Determine dose-limiting toxicities (DLTs) and maximum tolerated dose (MTD) of iv infusions of AsiDNA. | At Cycle 1 (a cycle is 21 days for Part A and 28 days for Part B) for all patients
  DLTs will be based on the toxicities observed during the first 3 weeks of study treatment (i.e, cycle 1: from Day 1 to Day 21) for Part A and during the 4 weeks of study treatment (i.e, cycle 1: from Day 1 to Day 28) for Part B.
  MTD is defined as the dose immediately below the unacceptable dose or defined as the highest tested dose if no DLT observed at this dose.

SECONDARY OUTCOMES:
Collection of new Adverse Events and follow-up of all ongoing Adverse Events assessed | At Cycle 1 (at Day 1; Day 3; Day 8; Day 15) and at Cycle 2 (at Day 1; Day 8; Day 15) and at each subsequent cycles in any (at Day 1; Day 8; Day 15) for all patients
  Adverse Events will be reported and graded based on the National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events (AE) [CTCAE] scale, version 4.03.
Elimination half-life (t1/2) of iv infusions of AsiDNA | At Cycle 1 (at Day 1; Day 3; Day 8; Day 15) and at cycle 2 (at Day 1) for all patients
  The following standard plasma PK parameter for IV AsiDNA will be analyzed:
  elimination half-life (t1/2) in hours
ECG evaluation for safety assessment | Before each cycle (e.g at Day 1 of cycle 1; Day 1 of cycle 2 and Day 1 of each subsequent cycles if any) per usual center's practice.
  12-lead ECG will be performed before each cycle (e.g at Day 1 of cycle 1; Day 1 of cycle 2 and Day 1 of each subsequent cycles if any) per usual center's practice.
Peak plasma concentration of iv infusions of AsiDNA | At Cycle 1 (at Day 1; Day 3; Day 8; Day 15) and at cycle 2 (at Day 1) for all patients
  The following standard plasma PK parameter for IV AsiDNA will be analyzed:
  peak plasma concentration (Cmax) in ng/mL
Time to peak plasma concentration of iv infusions of AsiDNA | At Cycle 1 (at Day 1; Day 3; Day 8; Day 15) and at cycle 2 (at Day 1) for all patients
  The following standard plasma PK parameter for IV AsiDNA will be analyzed:
  time to peak plasma concentration (tmax) in hours
Area under the curve of iv infusions of AsiDNA | At Cycle 1 (at Day 1; Day 3; Day 8; Day 15) and at cycle 2 (at Day 1) for all patients
  The following standard plasma PK parameter for IV AsiDNA will be analyzed:
  area under the curve (AUC) in mg*h/L.
Accumulation factor based on total plasma exposure of iv infusions of AsiDNA | At Cycle 1 (at Day 1) and at cycle 2 (at Day 1) for all patients
  The following standard plasma PK parameter for IV AsiDNA will be analyzed:
  accumulation factor between Day 1 and Day 3 based on total plasma exposure.

CONTACTS AND LOCATIONS:
Locations (5):
- Belgium (2):
  - Institut Jules Bordet, Brussels
  - Grand Hôpital de Charleroi, Charleroi
- France (3):
  - Centre Leon Berard, Lyon
  - Institut Curie, Paris
  - Institut Claudius Regaud, Toulouse

REFERENCES:
- [Derived] Le Tourneau C, Delord JP, Kotecki N, Borcoman E, Gomez-Roca C, Hescot S, Jungels C, Vincent-Salomon A, Cockenpot V, Eberst L, Mole A, Jdey W, Bono F, Trochon-Joseph V, Toussaint H, Zandanel C, Adamiec O, de Beaumont O, Cassier PA. A Phase 1 dose-escalation study to evaluate safety, pharmacokinetics and pharmacodynamics of AsiDNA, a first-in-class DNA repair inhibitor, administered intravenously in patients with advanced solid tumours. Br J Cancer. 2020 Nov;123(10):1481-1489. doi: 10.1038/s41416-020-01028-8. Epub 2020 Aug 25. PMID 32839491
- See also: Sponsor website — http://www.onxeo.com